CLINICAL TRIAL: NCT03724838
Title: Esomeprazole Alone or With Sildenafil Citrate in Women With Early-onset Preeclampsia: A Randomized Controlled Trial
Brief Title: Esomeprazole With Sildenafil Citrate in Women With Early-onset Preeclampsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: aswu 193/7/18
Record Dates: First submitted 2018-10-29; First posted 2018-10-30 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Preeclampsia
Keywords: Esomeprazole; Sildenafil Citrate; preterm preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Esomeprazole; Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: We will conduct a randomized, double-blind, placebo-controlled trial designed to evaluate the efficacy and safety of Esomeprazole alone or with Sildenafil Citrate in preterm pregnancies complicated by preeclampsia.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: both participants and researchers will be blinded to the intervention given
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Esomeprazole with Sildenafil Citrate (Active Comparator): Patients will take esomeprazole single dose of 40 mg orally once a day plus three doses of Sildenafil Citrate 40mg orally every 8 hours
  Interventions: Drug: Esomeprazole with Sildenafil Citrate; Drug: Sildenafil Citrate
- Esomeprazole alone plus placebo to Sildenafil Citrate (Active Comparator): Patients will take esomeprazole single dose of 40 mg orally once a day plus three doses of placebo identical in shape and consistency withSildenafil Citrate 40mg orally every 8 hours
  Interventions: Drug: Esomeprazole with Sildenafil Citrate; Drug: Placebo to Sildenafil Citrate
- placebo to Esomeprazole plus placebo to Sildenafil Citrate (Placebo Comparator): Patients will take placebo identical in shape and consistency with esomeprazole single dose of 40 mg orally once a day plus three doses of placebo identical in shape and consistency withSildenafil Citrate 40mg orally every 8 hours
  Interventions: Drug: Placebo to Esomeprazole; Drug: Placebo to Sildenafil Citrate

INTERVENTIONS:
Drug: Esomeprazole with Sildenafil Citrate — Patients will take esomeprazole single dose of 40 mg orally once a day
  Other Names: Active Comparator
  Arms: Esomeprazole alone plus placebo to Sildenafil Citrate; Esomeprazole with Sildenafil Citrate
Drug: Sildenafil Citrate — Patients will take Sildenafil Citrate 40mg every 8 hours
  Other Names: active comparator
  Arms: Esomeprazole with Sildenafil Citrate
Drug: Placebo to Esomeprazole — Patients will take inert tablets similar in appearance, color, and consistency to esomeprazole single dose of 40 mg orally once a day
  Arms: placebo to Esomeprazole plus placebo to Sildenafil Citrate
Drug: Placebo to Sildenafil Citrate — Patients will take inert tablets similar in appearance, color, and consistency to Sildenafil Citrate 40mg every 8 hours
  Arms: Esomeprazole alone plus placebo to Sildenafil Citrate; placebo to Esomeprazole plus placebo to Sildenafil Citrate

SUMMARY:
Previous studies have shown that expectant management of preeclampsia in the context of extreme prematurity may improve perinatal outcomes. Indeed, it has been estimated that for each additional day of pregnancy prolongation between 24 and 32 weeks of gestation, there is a nonlinear corresponding gain of 1% in fetal survival. In this study, we evaluate the use of Esomeprazole alone or with Sildenafil Citrate for the treatment of singleton pregnancies complicated by preeclampsia. We hypothesized that the potential increase in uteroplacental and fetoplacental blood flow with the use of Esomeprazole alone or with Sildenafil Citrate may be associated with pregnancy prolongation (the primary study outcome) and improved maternal and perinatal outcomes.

DETAILED DESCRIPTION:
The etiology and pathophysiology of preeclampsia have not been clearly established; impaired immunologic adaptation and genetic incompatibility seem to be involved in deficient trophoblastic implantation. Placental hypoxia and endothelial dysfunction may lead to preeclampsia through an exacerbated systemic inflammatory reaction. Increased placental expression and secretion of soluble fms-like tyrosine kinase 1 appear to play a central role in the pathogenesis of preeclampsia. The soluble fms-like tyrosine kinase 1 antagonizes the proangiogenic biologic activity of circulating vascular endothelial growth factor and placental growth factor, leading to a failure of nitric oxide signaling to smooth muscle The investigators will conduct a randomized, double-blind, placebo-controlled trial designed to evaluate the efficacy and safety of Esomeprazole alone or with Sildenafil Citrate in preterm pregnancies complicated by preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women presenting at a Gestational age between 28 + 0 weeks and 32 + 0 weeks presented with preterm preeclampsia
* The patient will be managed with an expectant management
* Give written informed consent

Exclusion Criteria:

* Multiple pregnancies.
* Previous hypersensitivity reaction esomeprazole or sildenafil citrate
* Contraindications to the use of esomeprazole or sildenafil citrate
* The patient is unable or unwilling to give consent
* An established fetal compromise that necessitates delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women with early-onset preeclampsia
Enrollment: 180 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Prolongation of gestation measured from the time of enrollment to the time of delivery. | 3 weeks
  Prolongation of gestation measured from the time of enrollment to the time of delivery

SECONDARY OUTCOMES:
Severe morbidity | 4 weeks
  Severe morbidity including eclampsia, liver or renal failure, hemolysis, elevated liver enzymes and low platelets syndrome (HELLP), disseminated intravascular coagulation (DIC), stroke, and pulmonary edema
Side effects | 4 weeks
  any side effects or adverse events related to the intervention, intervention stopped due to side effects
The change in serum level of sFlt-1 and endoglin before the start of treatment and at termination of pregnancy | 4 weeks
  The change in serum level of sFlt-1 and endoglin before the start of treatment and at termination of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No